CLINICAL TRIAL: NCT06549621
Title: Cardiotoxicity of Carbon Monoxide in Patients Treated With Hyperbaric Oxygen Therapy
Acronym: COCARDIOTOX
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: COCARDIOTOX (29BRC22.0049)
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Carbon Monoxide Poisoning
Keywords: cardiac injury; cardiac toxicity
MeSH Terms: conditions — Carbon Monoxide Poisoning; Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Carbon monoxide poisoning is a frequent domestic accident and the leading cause of death from unintentionnal poisoning. Its toxicity is based on the CO binding to hemoglobin and myoglobin, inhibition of mitochondrial cytochrome oxidase, resulting in tissue hypoxia and reduced adenosine triphosphate synthesis and ischemia-reperfusion injury.

This study aims to investigate the early and late cardiologic effects of CO in patients treated with hyperbaric oxygen (HBOT) for CO poisoning

DETAILED DESCRIPTION:
This is a single-center retrospective study on health data. The methodology includes a collection of data on health and history data of patients treated by HBOT fo CO poisoning between 01/01/2015 and 31/12/2021 and carrying out a telephone interview of patients who have had early cardiovascular manifestations of CO poisoning.

One month between the start of theses interviews, an information letter on the study is sent by post, giving the possibility of opposing it.

ELIGIBILITY:
Inclusion Criteria:

Patients treated for CO poisoning with HBOT in the hyperbaric and underwater medicine department of the Brest University hospital from 2015/01/01 to 2021/12/31

Exclusion Criteria:

* refusal

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients treated for CO poisoning with HBOT following European and French recommendations in our department from 2015/01/01 to 2021/12/31
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2024-10-25 (Estimated)

PRIMARY OUTCOMES:
early and late cardiac injury due to CO poisoning description | enrollment (inclusion)
  clinical manifestation, troponin elevation and/or ECG abnormality during acute CO poisoning description; then late cardiac manifestation and abnormality declared by patients who have had early cardiac abnormality (troponin elevation and/or ECG abnormalities)

SECONDARY OUTCOMES:
relationship between the source of CO poisoning and cardiac injury | enrollment (inclusion)
  comparison between the group of patients with early cardiac abnormalities (troponin elevation and/or ECG abnormalities) and the group of patients without early cardiac abnormalities using Ficher test
relationship between context of poisoning (domestic, professionnal or intentional poisoning) and cardiac injury | enrollment (inclusion)
  comparison between the group of patients with early cardiac abnormalities (troponin elevation and/or ECG abnormalities) and the group of patients without early cardiac abnormalities using Ficher test
relationship between other possibly associated poisoning and cardiac injury | enrollment (inclusion)
  comparison between the group of patients with early cardiac abnormalities (troponin elevation and/or ECG abnormalities) and the group of patients without early cardiac abnormalities using Ficher test
relationship between severity of neurological symptoms and cardiac injury | enrollment (inclusion)
  comparison between the group of patients with early cardiac abnormalities (troponin elevation and/or ECG abnormalities) and the group of patients without early cardiac abnormalities using Ficher test
relationship between cardiovascular risk factors or preexisting cardio vascular abnormality and cardiac injury | enrollment (inclusion)
  comparison between the group of patients with early cardiac abnormalities (troponin elevation and/or ECG abnormalities) and the group of patients without early cardiac abnormalities using Ficher test

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France